CLINICAL TRIAL: NCT00287443
Title: Metabolic Abnormalities in Hispanic Children With Cystic Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer with the University
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0303-161
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glucose Tolerance Test; Calorimetry, Indirect; Absorptiometry, Photon

INTERVENTIONS:
Procedure: Oral Glucose tolerance test
Procedure: Whole body protein turnover
Procedure: IV glucose tolerance test
Procedure: Indirect Calorimetry
Procedure: Dual Energy X-ray Absorptiometry (DEXA)
Procedure: Growth Hormone Stimulation Test

SUMMARY:
Our specific aims include:

1. AIM 1. Characterization of glucose tolerance, nutritional and clinical status, socioeconomic status, family history of diabetes and genotype in Hispanic CF children compared to Caucasian CF children. Each child will undergo a two-hour oral glucose tolerance test and will be categorized by glucose tolerance according to standards set forth by the 1998 CF Consensus Conference on Diabetes. Nutritional status will be determined by three-day food journals and intake will be compared to energy needs measured by indirect calorimetry. Socio-economic status will be calculated from reported family income and medical insurance coverage. Genotyping will be done at the laboratory of Dr. Arthur Beaudet at Baylor College of Medicine. Clinical status will be measured using modified NIH scores. Family history for both type 1 and type 2 diabetes will be obtained in Spanish by Dr.Vanderwel. This specific aim tests the hypothesis that glucose intolerance /frank CF related diabetes occurs at a younger age in Hispanics than in Caucasians with CF, and is correlated to family history of diabetes and clinical status.
2. AIM 2. Characterization of insulin secretion and insulin sensitivity. Previous studies in adults have described peripheral insulin resistance as a major cause of CF related diabetes, yet studies have not been conducted in children. Studies in adults and children without CF suggest that insulin resistance occurs more frequently in Hispanics. We will measure insulin secretion and insulin sensitivity using the frequently sampled intravenous glucose tolerance test (IVGTT) and the minimal model analysis of Bergman, as modified for children. This specific aim tests the hypothesis that Hispanic children with CF have worse peripheral insulin resistance, but similar insulin secretion when compared to Caucasian children with CF.
3. AIM 3. Quantification of post-absorptive gluconeogenesis and whole body protein turnover. Total hepatic glucose production (HGP) will be measured using [6,6-2H2]glucose. We will quantify gluconeogenesis by measurement of the incorporation of 2H into the 2nd, 5th and 6th carbons of glucose following 2H20 administration method of Landau). We will determine whole body protein turnover using the stable isotopes [1-13C]leucine and will measure serum amino acid levels. This specific aim tests the hypothesis that gluconeogenesis and whole body protein turnover are disproportionately higher in Hispanic children and adolescents with CF than in Caucasian CF children.

DETAILED DESCRIPTION:
We will recruit 12 Hispanic prepubertal children with CF (ages 7-12, Tanner I) and 12 Hispanic adolescents (ages 15-17, Tanner 3 or 4) from the CF Centers at University of Texas Southwestern and Baylor College of Medicine in Houston. Information obtained from these subjects will be compared to 12 prepubertal and 12 adolescent Caucasian children with CF recruited from the same CF centers. We will categorize the subjects according to glucose tolerance (OGTT), as well as insulin secretion and insulin sensitivity using the IVGTT and the Minimal Model, as modified for children. We will also compare the historical information of socio-economic status and family history. Clinical status will be characterized by measuring pulmonary function and modified NIH scores, in addition to measuring levels of circulating cytokines. Gluconeogenesis (GNG) will be quantified by measuring the incorporation 2H into the 2nd, 5th and 6th carbons of glucose. Whole body protein turnover (WBPT) will be measured using [1-13C]leucine. Nutritional status will be determined by three-day food journals, and intake will be compared to energy needs, utilizing indirect calorimetry to measure resting energy expenditure. Subjects will be recruited from the CF centers at the University of Texas- Southwestern and the South Central CF Consortium.

ELIGIBILITY:
Inclusion Criteria: Subjects will be required to be medically stable at the time of the study. Medical stability will be defined as:

1. No hospital admission for six weeks or more before the study
2. No oral or intravenous antibiotics for at least six weeks preceding the study (subjects will be allowed to use low doses of inhaled corticosteroids)
3. Weight-stable (weight deviation less than 2.5 kilograms) for two months prior to the study.

Exclusion Criteria:

1. Use of oral or intravenous corticosteroid medications within six weeks of the study
2. Evidence of severe liver disease (hepatomegaly, 30% or greater elevation of liver transaminases, listed for liver transplant)
3. Colonization with Burkholderia cepacia
4. Pregnancy
5. Patients requiring supplemental oxygen.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-02-02 (Estimated); Primary Completion 2006-02-02 (Estimated); Study Completion 2006-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana s HArdin, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- Children's Medical Center of Dallas, Dallas, Texas, United States